CLINICAL TRIAL: NCT02928783
Title: Evaluation of Exercise Tolerance and Cardiac Output in Patients With Heart Failure After Intervention of Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Jin Long Huang, M.D., P.D, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CG13107
Record Dates: First submitted 2016-09-04; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure With or Without CRT-P/D
Keywords: Home-based cardiac rehabilitation; Quality of Medical Care; Heart Failure
MeSH Terms: conditions — Heart Failure

ARMS (2):
- Intervention (Experimental): In interventional group, we arranged individualized rehabilitation programs including home-based cardiac rehabilitation, diet education and management of daily activity for 3 months.
  Interventions: Behavioral: Home-based cardiac rehabilitation
- Control (No Intervention): We didn't arrange individualized rehabilitation programs including home-based cardiac rehabilitation, diet education and management of daily activity for 3 months.

INTERVENTIONS:
Behavioral: Home-based cardiac rehabilitation
  Arms: Intervention

SUMMARY:
Home-based rehabilitation programs have not been widely few been studied and the training effects are not unclear. This study evaluates the beneﬁcial effects of home-based cardiac rehabilitation on quality of medical care in patients with chronic heart failure.

DETAILED DESCRIPTION:
cardiopulmonary rehabilitation programs are safe and effective for improving functional capacity, quality of life, as well as for reducing in the re-admission rate and all-cause mortality of patients with heart failure.clinical trials that have established the benefits of hospital-based cardiac rehabilitation for patients with chronic heart failure. Home-based cardiac rehabilitation could be more accessible and acceptable compared with hospital-based cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with NYHA I, II, III, and LVEF<50%.

Exclusion Criteria:

* Heart failure patients with NYHA I, II, III, and LVEF<50%. But excluded pregnancy, disability.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline peak oxygen uptake (ml /kg/min) at 3 months | 3 months
  All participants the assessment of cardiopulmonary exercise test at baseline and after completing an 3 months training programs.
Change from Baseline quality of life at 3 months | 3 months
  All participants the assessment of Minnesota Living With HF Questionnaire (MLHFQ) at baseline and after completing an 3 months training programs.
Change from Baseline 6-min walking distance (6MWD) at 3 months | 3 months
  All participants the assessment of 6-min walk test at baseline and after completing an 3 months training programs.

SECONDARY OUTCOMES:
readmission rate | 90 days
  All participants the assessment of 90-day readmission rate after completing an 3 months training programs.

REFERENCES:
- [Result] Haykowsky MJ, Liang Y, Pechter D, Jones LW, McAlister FA, Clark AM. A meta-analysis of the effect of exercise training on left ventricular remodeling in heart failure patients: the benefit depends on the type of training performed. J Am Coll Cardiol. 2007 Jun 19;49(24):2329-36. doi: 10.1016/j.jacc.2007.02.055. Epub 2007 Jun 4. PMID 17572248
- [Result] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Result] Tomczak CR, Thompson RB, Paterson I, Schulte F, Cheng-Baron J, Haennel RG, Haykowsky MJ. Effect of acute high-intensity interval exercise on postexercise biventricular function in mild heart failure. J Appl Physiol (1985). 2011 Feb;110(2):398-406. doi: 10.1152/japplphysiol.01114.2010. Epub 2010 Nov 18. PMID 21088202
- [Result] Smart NA, Steele M. A comparison of 16 weeks of continuous vs intermittent exercise training in chronic heart failure patients. Congest Heart Fail. 2012 Jul-Aug;18(4):205-11. doi: 10.1111/j.1751-7133.2011.00274.x. Epub 2011 Nov 27. PMID 22809258
- [Result] Schmidt C, Theilmeier G, Van Aken H, Korsmeier P, Wirtz SP, Berendes E, Hoffmeier A, Meissner A. Comparison of electrical velocimetry and transoesophageal Doppler echocardiography for measuring stroke volume and cardiac output. Br J Anaesth. 2005 Nov;95(5):603-10. doi: 10.1093/bja/aei224. Epub 2005 Sep 9. PMID 16155037
- [Result] Suttner S, Schollhorn T, Boldt J, Mayer J, Rohm KD, Lang K, Piper SN. Noninvasive assessment of cardiac output using thoracic electrical bioimpedance in hemodynamically stable and unstable patients after cardiac surgery: a comparison with pulmonary artery thermodilution. Intensive Care Med. 2006 Dec;32(12):2053-8. doi: 10.1007/s00134-006-0409-x. Epub 2006 Oct 13. PMID 17039348 (Retraction: PMID 21604011 Intensive Care Med. 2011 Jul;37(7):1232)